CLINICAL TRIAL: NCT01750294
Title: A Pilot Study of Chlorthalidone Among Patients With Poorly Controlled Hypertension and CKD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1206009002; 1206009002 (Other: IRB)
Record Dates: First submitted 2012-12-12; First posted 2012-12-17 (Estimated); Results first posted 2016-05-10 (Estimated); Last update posted 2016-06-13 (Estimated); Status verified 2016-05

CONDITIONS: Chronic Kidney Disease; Poorly-Controlled Hypertension
Keywords: hypertension; kidney disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hypertension; Kidney Diseases | interventions — Chlorthalidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Chlorthalidone

SUMMARY:
It is estimated that in the United States there are approximately 8 million individuals with moderate to severe chronic kidney disease (CKD), not on dialysis. Volume expansion plays an important role in the pathogenesis of hypertension in patients with CKD. For this pilot study, the investigators hypothesize that administration of chlorthalidone among patients with moderate to severe CKD will improve blood pressure (BP).

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years.
* Estimated glomerular filtration rate (eGFR) ≤ 45 ml/min/1.73m2 but ≥20 mL/min/1.73m2.
* Poorly controlled blood pressure by 24-hour ambulatory blood pressure (BP) monitoring.
* Treated hypertension: use of at least one antihypertensive drug. One of the drugs should be either an angiotensin converting enzyme (ACE) inhibitor or angiotensin receptor blocker (ARB). If these are contraindicated then use of a beta-blocker is required.

Exclusion Criteria:

* Use of thiazide or thiazide-like drugs in the previous 3 months.
* Use of furosemide in a dose >200 mg/d.
* Ambulatory BP of either ≥160 systolic or ≥100 mmHg by 24-hour ambulatory BP monitoring.
* Expected to receive renal replacement therapy within the next 3 months.
* Vascular event such as myocardial infarction, heart failure hospitalization, or stroke within 3 months prior to randomization.
* Pregnant or breastfeeding women or women who are planning to become pregnant or those not using a reliable form of contraception (oral contraceptives. condoms and diaphragms will be considered reliable).
* Known hypersensitivity to thiazide or sulfa drugs.
* Organ transplant recipient or therapy with immunosuppressive agents. Nasal or inhaled corticosteroids will be permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-08; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rajiv Agarwal, MD FASN FAHA, Principal Investigator — Indiana University
Locations (1):
- Richard L. Roudebush VAMC, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the VA Medical Center from Sept. 18, 2012 - May 15, 2013. Eligible subjects were ≥ 18 years of age with estimated glomerular filtration rate ≤ 45 but > 20 mL/min/1.73m2. The study initially recruited subjects with resistant hypertension but was amended to include those with poorly controlled but treated hypertension.
Pre-assignment Details: Prior to assignment, participants completed home blood pressure monitoring, ambulatory blood pressure monitoring, and a two-week run-in period, during which all subjects received a standard anti-hypertensive regimen based on the existing regimen of the subject.
Groups:
- Chlorthalidone: Open-label, forced-titration of Chlorthalidone (25mg/day at baseline)
Period: Overall Study
Arm/Group | Chlorthalidone
Started | 14
Completed | 12
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Safety Endpoint | 1

BASELINE CHARACTERISTICS:
Population: Participants who completed the two-week run-in and enrolled in the study are included in the baseline analysis.
Arm/Group | Chlorthalidone
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.5 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Chronic Kidney Disease (CKD) Stage [Number; unit: participants] — Staging captured according to estimated glomerular filtration rate (eGFR) at baseline using the National Kidney Foundation (NKF) Kidney Disease Outcomes Quality Initiative (KDOQI) guidelines for staging chronic kidney disease (CKD).
  participants
    Stage 3B | 4
    Stage 4 | 8
    Stage 5 | 2
Estimated GFR [Mean (Standard Deviation); unit: mL/min/1.73m2] — Measured after two-week run-in
  mL/min/1.73m2 | 26.8 (8.8)

OUTCOME MEASURES:

1. Primary Outcome: Change of Systolic Ambulatory Blood Pressure From Baseline to 12 Weeks
Time Frame: Baseline and 12 weeks after intervention
Population: Intention to treat analysis (includes completers and non-completers)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Chlorthalidone
Number analyzed (Participants) | 14
mmHg | -10.5 (4.2)
Statistical Analysis 1: Comparison: Chlorthalidone; Test type: Superiority or Other; p = 0.01, Mixed Models Analysis — a = 0.05

ADVERSE EVENTS:
Time Frame: Baseline (week 0) through study completion (week 12)
Arm/Group | Chlorthalidone
Serious Adverse Events (participants affected / at risk) | 2/14
Other Adverse Events (participants affected / at risk) | 7/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chlorthalidone (N=14)
Elective kidney biopsy (Renal and urinary disorders) | 1 (1) — Subject experienced a drop in hemoglobin following an elective kidney biopsy and was admitted for concern of internal bleeding, which was absent on a computerized tomography (CT) scan.
New-onset ischemic stroke (Nervous system disorders) | 1 (1) — Occurred in a subject with a history of strokes, seizures, and co-morbid diabetes mellitus who volitionally stopped all anti-hypertensive medications.
Hypotension (Vascular disorders) | 1 (2) — Occurred in a subject with a history of strokes, seizures, and co-morbid diabetes mellitus who volitionally stopped all anti-hypertensive medications.
Syncope (Nervous system disorders) | 1 (2) — Occurred in a subject with a history of strokes, seizures, and co-morbid diabetes mellitus who volitionally stopped all anti-hypertensive medications.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chlorthalidone (N=14)
Hypokalemia (Metabolism and nutrition disorders) | 4 (4)
Hyperuricemia (Metabolism and nutrition disorders) | 4 (4)
Hyponatremia (Metabolism and nutrition disorders) | 3 (3)
Transient elevations of serum creatinine (Investigations) | 3 (3)
Dizziness (Nervous system disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No